CLINICAL TRIAL: NCT06823778
Title: Prophylactic Radiofrequency Left Atrial Posterior Wall Isolation (box Lesion Ablation) to Prevent Atrial Fibrillation After Cardiac Surgery (PROBOX): a Randomized Controlled Trial
Brief Title: Prophylactic Radiofrequency Left Atrial Posterior Wall Isolation to Prevent Atrial Fibrillation After Cardiac Surgery
Acronym: PROBOX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vasily I. Kaleda (Other)
Responsible Party: Sponsor-Investigator, Vasily I. Kaleda, Principal Investigator, Yudin Hospital
Organization: Yudin Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1.2025
Record Dates: First submitted 2025-02-02; First posted 2025-02-12 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Atrial Fibrillation
Keywords: Postoperative Atrial Fibrillation; Radiofrequency Ablation; Box Lesion Ablation; Prophylactic Ablation
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: A Prospective Parallel-Arm Single-Blind Randomized Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (No Intervention): No ablation will be performed in this group of patients.
- Intervention (Experimental): In this group of patients, radiofrequency left atrial posterior wall isolation will be performed.
  Interventions: Device: Radiofrequency ablation

INTERVENTIONS:
Device: Radiofrequency ablation — In this group of patients, epicardial radiofrequency left atrial posterior wall isolation will be performed with AtriCure Isolator Synergy OLL2 bipolar radiofrequency clamp without opening the left atrium.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to learn if an epicardial radiofrequency left atrial posterior wall isolation (box lesion ablation) prevents atrial fibrillation after cardiac surgery. The main question it aims to answer is:

- Does box lesion ablation lower the number of patients experiencing de-novo atrial fibrillation requiring any treatment after cardiac surgery? Researchers will compare box lesion ablation to no ablation to see if ablation prevents postoperative atrial fibrillation.

Participants will undergo ablation or no ablation at the time of other cardiac surgery.

Data will be collected while in hospital. Additional information will be collected on 30th day after surgery by telephone call or during a visit.

DETAILED DESCRIPTION:
Postoperative atrial fibrillation (POAF) is a common complication after heart surgery that occurs in 10-60% of patients. It can cause hypotension, tachycardia, stroke, systemic embolism, or heart failure, and is associated with increased mortality rates, prolonged hospital stays and increased costs. Several studies have investigated the use of radiofrequency ablation (the standard of surgical care for atrial fibrillation during concomitant cardiac surgery when the diagnosis is known preoperatively) to prevent POAF. However, these studies were limited mainly to pulmonary vein isolation and had methodological limitations such as small sample sizes, inclusion/exclusion criteria, and randomization procedures, and have not translated into clinical practice changes. The current study aims to investigate the use of radiofrequency left atrial posterior wall isolation, also known as box lesion ablation, as a more effective treatment compared to pulmonary vein isolation, in a properly designed randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing cardiac surgery by a single surgeon (V.K.)
* Informed consent

Exclusion Criteria:

* History of atrial fibrillation/flutter
* Minimally invasive approach
* Off-pump surgery
* Emergent/salvage surgery
* Severe pericardial adhesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative Atrial Fibrillation | Within 30-day of surgery or until discharge, whichever came last, assessed up to 6 months after surgery
  Incidence of clinically significant (requiring any type of intervention) postoperative atrial fibrillation

SECONDARY OUTCOMES:
Postoperative Mortality | Within 30-day of surgery or until discharge, whichever came last, assessed up to 6 months after surgery
  All deaths occurring during the hospitalization in which the operation was performed, even if after 30 days; and all deaths occurring after discharge from the hospital, but before the end of the 30th postoperative day.
Postoperative Stroke | Within 30-day of surgery or until discharge, whichever came last, assessed up to 6 months after surgery
  Number of patients who have a postoperative stroke (i.e., any confirmed neurological deficit of abrupt onset caused by a disturbance in blood supply to the brain) that did not resolve within 24 hours
Length of Stay | Up to 6 months after surgery
  Postoperative length of in-hospital stay
Unplanned Readmission | Within 30 days after surgery
  Unplanned 30-day any cause readmission rate

OTHER OUTCOMES:
Operative time | Up to 24 hours after the start of the operation
  Total operative time (min)
Cardiopulmonary bypass time | Up to 24 hours after the start of the operation
  Total cardiopulmonary bypass time (min)
Cross-clamp time | Up to 24 hours after the start of the operation
  Total cross-clamp time (min)
Other arrhythmias rate | Within 30-day of surgery or until discharge, whichever came last, assessed up to 6 months after surgery
  Any arrhytmias other than POAF rate

CONTACTS AND LOCATIONS:
Overall Officials: Alexandr Piskun, M.D., Ph.D., Study Chair — Yudin Hospital
Locations (1):
- Department of Cardiac Surgery, Yudin Hospital, Moscow, Moscow, Russia

REFERENCES:
- [Background] Visanji M, Belley-Cote EP, Pandey A, Amit Y, McClure GR, Young J, Um KJ, Oraii A, Healey JS, Whitlock RP, McIntyre WF. Prophylactic ablation during cardiac surgery in patients without atrial fibrillation: a systematic review and meta-analysis of randomized trials. Interdiscip Cardiovasc Thorac Surg. 2024 Dec 3;39(6):ivae195. doi: 10.1093/icvts/ivae195. PMID 39589863
- [Background] Kaleda VI, Snegirev MA, Efendiev VU, Piskun AV, Batukov IA, Nazaryan KE, Pidanov OY. Concomitant Box Lesion Ablation for Atrial Fibrillation with a Standard Non-Irrigated Bipolar Radiofrequency Clamp: Simplified Approach Without Left Atriotomy. Braz J Cardiovasc Surg. 2025 Feb 17;40(2):e20230432. doi: 10.21470/1678-9741-2023-0432. PMID 39960384